CLINICAL TRIAL: NCT06453317
Title: Comparison of Ustekinumab, Infliximab and Combination Therapy in Moderately to Severely Active Ulcerative Colitis (COMBO-UC)
Brief Title: Comparison of Ustekinumab, Infliximab and Combination Therapy in Moderately to Severely Active Ulcerative Colitis
Acronym: COMBO-UC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of Lodz (Other)
Collaborators: Poznan University of Medical Sciences (Other); Clinical Hospital Heliodor Swiecicki of the Medical University of Karol Marcinkowski in Poznań (Other); Norbert Barlicki Memorial Teaching Hospital No. 1 of the Medical University of Lodz (Unknown); Medical Research Agency, Poland (Other Government)
Responsible Party: Principal Investigator, Renata Talar-Wojnarowska, Principal Investigator, Medical University of Lodz
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Combo/2022/3; 2023-506452-25 (EudraCT Number)
Record Dates: First submitted 2024-05-24; First posted 2024-06-11 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2024-11

CONDITIONS: Ulcerative Colitis; Inflammatory Bowel Diseases
Keywords: dual biological therapy; infliximab; ustekinumab; Inflammatory Bowel Diseases; Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases | interventions — Infliximab; Ustekinumab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Due to the comparative nature of the study, aiming to compare the effectiveness of dual biological therapy with biologic drugs administered solely, we have not implemented treatment blinding. However, a blinded central endoscopy reader was included. Each endoscopy procedure will be recorded using an external device and sent to the central reader who will be blinded to the patient's treatment arm. It is important to note that the final decision regarding the endoscopic disease activity will remain with the endoscopist performing the procedure.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Infliximab (Active Comparator): Infliximab 5 mg/kg i.v at Weeks 0, 2, 6 and then every 8 weeks for 52 weeks.
  Interventions: Biological: Infliximab
- Ustekinumab (Active Comparator): Ustekinumab: first dose i.v. at Week 0 (Patients with body weight ≤55 kg - 260 mg, patients with body weight >55-≤85 kg 390 mg, patients with body weight >85 kg - 520 mg) then 90 mg s.c. every 8/12 weeks for 52 weeks.
  Interventions: Biological: Ustekinumab
- Infliximab + Ustekinumab (Experimental): Infliximab 5 mg/kg i.v. at Week 0, 2, 6.
  + Ustekinumab: first dose i.v. at Week 0 (Patients with body weight ≤55 kg - 260 mg, patients with body weight >55-≤85 kg 390 mg, patients with body weight >85 kg - 520 mg) then 90 mg s.c. every 8/12 weeks for 52 weeks
  Interventions: Biological: Infliximab; Biological: Ustekinumab

INTERVENTIONS:
Biological: Infliximab — Infliximab 5 mg/kg i.v at Weeks 0, 2, 6 and then every 8 weeks for 52 weeks.
  Arms: Infliximab; Infliximab + Ustekinumab
Biological: Ustekinumab — Ustekinumab: first dose i.v. at Week 0 (Patients with body weight ≤55 kg - 260 mg, patients with body weight >55-≤85 kg 390 mg, patients with body weight >85 kg - 520 mg) then 90 mg s.c. every 8/12 weeks for 52 weeks.
  Arms: Infliximab + Ustekinumab; Ustekinumab

SUMMARY:
The goal of this clinical trial is to learn if combined therapy with infliximab and ustekinumab works better than using these drugs alone in adult patients with ulcerative colitis. It will also learn about the safety of this combination. The main questions it aims to answer are:

Does the combination therapy improve the symptoms and heal the intestine quicker and better than these drugs administered alone? Does the combination therapy improve the quality of life better than these drugs administered alone? What medical problems do participants have when taking the combination therapy?

Participants:

Patients diagnosed with UC will be qualified to biologic therapy (infliximab/ustekinumab/infliximab + ustekinumab).

Visit the clinic in stated periods for assessment and to apply medication. Take drugs based on the schedule.

ELIGIBILITY:
Inclusion Criteria:

1. Obtaining informed, written consent for the patient's participation in the in the study and for all planned procedures.
2. Age ≥ 18 years and ≤65 at the time of screening.
3. In the case of women of reproductive potential, agreement to not donate oocytes for the entire period of participation in the in the study and 6 months after receiving the last dose of the drug.
4. For women of reproductive potential, agreement to use effective contraception (Table 4) during the entire period, during which the patient participates in the study and for a period counted from the last dose of 15 weeks if using UST (patients in arms B and C) or 6 months if using IFX (patients in arm A).
5. Negative serum or urine pregnancy test in women of childbearing age.
6. Diagnosis of UC a minimum of. 3 months prior to screening documented by:

   (a) medical source documentation of the patient with the result of an endoscopic examination that diagnosed features typical of UC.

   (b) a histopathological examination result consistent with UC. In the absence of a histopathological result, it is possible to take sections during the endoscopic examination for histopathological evaluation at the time of eligibility for the study with subsequent sending of the material to the local pathomorphology laboratory to confirm the diagnosis of UC before randomization.
7. UC with moderate or severe activity defined as a Mayo scale score (Appendix 2) of 7 to 12 including the following sub-item values (each sub-item 0-3 points depending on the severity of the lesions):

   - Frequency of bowel movements
   * Bowel bleeding
   * Endoscopic image of the colonic mucosa
   * General medical evaluation and:
   * with inadequate response to standard treatment, including corticosteroids and 6-mercaptopurine or azathioprine, or.
   * intolerant of treatment with corticosteroids and 6-mercaptopurine or azathioprine, or
   * having contraindications to treatment with corticosteroids and 6-mercaptopurine or azathioprine, or
   * with loss of response to standard treatment, including to treatment with corticosteroids and 6-mercaptopurine or azathioprine, including patients:
   * Steroid-resistant - in whom there is no clinical improvement despite the use of a daily steroid up to 0.75 mg/kg prednisolone for 4 weeks;
   * Steroid-dependent - in whom failure to reduce the steroid dose below 10 mg/day, converted to prednisolone, within 3 months of starting steroid therapy or relapse of complaints within 3 months of steroid withdrawal.
   * Refractory patients/about inadequate response to immunosuppressive treatment, defined as lack of remission or recurrence of complaints despite immunosuppressive treatment for at least 3 months at appropriate doses (azathioprine 2-2.5 mg/kg/day or 6-mercaptopurine 1-1.5 mg/kg/day).
8. Patients taking 5-ASA derivatives, corticosteroids, immunosuppressants may be included in the study if they are taking a fixed and specified dose of the above drugs 14 days before the day of randomization.

Exclusion Criteria:

1. Previous use of the study drug IFX or UST.
2. Hypersensitivity to the active substance or excipients.
3. Moderate or severe myocardial insufficiency (NYHA III or IV).
4. Unstable coronary artery disease.
5. History of serious cerebrovascular disease (stroke, intracranial hemorrhage, transient cerebral ischemia) within the last 24 weeks prior to screening.
6. Chronic respiratory failure.
7. Severe chronic renal failure.
8. Severe chronic liver failure.
9. Demyelinating syndrome or symptoms resembling the syndrome.
10. Alcoholic disease, post-alcoholic liver damage.
11. Diagnosis of malignant neoplasms, including within 5 years preceding the time of eligibility for the program (except for carcinoma in situ of the cervix, and non-melanoma skin cancers).

12 Complications requiring other management (e.g., surgery). 13. Current or recent (defined as an incident within 12 weeks prior to randomization) documented episode of fulminant colitis, or intra-abdominal abscess, or acute colonic distension, or bowel perforation.

14. Status after extensive colorectal resection, subtotal or total colectomy with or without colostomy, or J-pouch reservoir.

15. Indication of surgical intervention due to underlying disease or when there is a suspicion of need for such intervention during the course of the study.

16. History of current or previously documented unclassified colitis or ischemic colitis.

17. History of colonic diverticulitis within the last 60 days prior to the randomization visit.

18. Current adenomatous polyps of the colon, small- or large-grade dysplasia in colon specimens, or previously diagnosed foci of large-grade dysplasia that have not been treated.

19. Enteral nutrition or total parenteral nutrition. 20. Pregnancy or breastfeeding. 21. Taking medications on the prohibited drugs list (Section 7.4.6). 22. daily dose of prednisone> 40 mg (or equivalent other corticosteroid) or budesonide MMX > 9 mg.

23. Status after bone marrow transplantation. 24. Condition after apheresis 12 months prior to the randomization visit. 25. Period after administration of allowed biologic drugs shorter than the drug's washout period from the body (Section 7.2).

26. Period after intestinal microbiota transplantation less than 8 weeks before signing informed consent to participate in the study.

27. Active or latent form of tuberculosis. 28. HIV infection. 29. Treatment period for active lesions of chronic infections (including pneumocystodosis, CMV, HPV, HSV infection, atypical mycobacteriosis, invasive bacterial or fungal infections).

30 History of HSV, HPV, influenza virus, SARS-CoV2 infection within 12 weeks prior to randomization or history of disseminated or complicated HSV infection.

31. History of congenital or acquired immunodeficiency. 32. receipt of live vaccine within 30 days prior to randomization. 33. infection with HBV or HCV. 34. Clinically significant changes on chest X-ray or ECG. 35 Clinically significant changes observed in laboratory test results:

1. ALT activity >3x the upper limit of normal (GGN)
2. AST activity >3x GGN
3. Total bilirubin level >2x GGN (exception is Gilbert syndrome when other causes of isolated hyperbilirubinemia are excluded).
4. ALP or GGTP activity >3x GGN
5. Creatinine level >2x GGN or impaired renal function (eGFR) <45mL/min calculated by MDRD formula.
6. Hemoglobin level <9g/dL
7. Absolute leukocyte count <3000/mm3
8. Absolute lymphocyte count <750/mm3
9. Neutrophil level <1000/mm3
10. Platelet level <100000/mm3. 36. Positive stool culture for bacteria/fungus (if clinically relevant in the opinion of the investigator).

    37.Positive stool culture for Clostridioides difficile. 38. Use of treatment not permitted under this protocol.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 172 (Estimated)
Dates: Start 2025-02-17 (Actual); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with clinical and endoscopic remission after the induction phase. | Week 14 for Infliximab arm and Week 16 for Ustekinumab and Infliximab + Ustekinumab arms
  Clinical remission: PRO-2 score ≤1 points, total Mayo score <3 Endoscopic remission: endoscopic Mayo score ≤1

SECONDARY OUTCOMES:
Percentage of patients with clinical response after the induction phase. | Week 14 for Infliximab arm and Week 16 for Ustekinumab and Infliximab + Ustekinumab arms
  Clinical response: change in PRO-2 score ≥50% or a change in total Mayo score ≥3 points
Percentage of patients with clinical response at Week 52. | Week 52
  Clinical response: change in PRO-2 score ≥50% or a change in total Mayo score ≥3 points
Percentage of patients with clinical remission at Week 52. | Week 52
  Clinical remission: PRO-2 score ≤1 points, total Mayo score <3
Percentage of patients with endoscopic response or remission after the induction phase and at Week 52 | Week 14 for Infliximab arm and Week 16 for Ustekinumab and Infliximab + Ustekinumab arms and Week 52
  Endoscopic response: change in endoscopic Mayo score ≥1 point Endoscopic remission: endoscopic Mayo score ≤1
Percentage of patients with biochemical remission after the induction phase and at Week 52. | Week 14 for Infliximab arm and Week 16 for Ustekinumab and Infliximab + Ustekinumab arms and Week 52
  Biochemical remission: calprotectin level ≤125 µg/g of stool
Percentage of patients with histological remission after the induction phase. | Week 14 for Infliximab arm and Week 16 for Ustekinumab and Infliximab + Ustekinumab arms
  Deep remission: PRO-2 score = 0 points, endoscopic Mayo score = 0 points and Picasso Histologic Remission Index = 0 points
Comparison of patients' quality of life after the induction phase and at Week 52 using 36-Item Short Form Survey (SF-36) and Inflammatory Bowel Disease Questionnaire (IBDQ). | Week 14 for Infliximab arm and Week 16 for Ustekinumab and Infliximab + Ustekinumab arms and Week 52
  SF-36: 0-100 points (a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability).
  IBDQ: 32-224 points (higher scores representing better quality of life).
Comparison of incidence of treatment-emergent adverse events after the induction phase and at Week 52. | Week 14 for Infliximab arm and Week 16 for Ustekinumab and Infliximab + Ustekinumab arms and Week 52
  Treatment-emergent adverse events and serious adverse events will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Renata Talar-Wojnarowska, Prof., Principal Investigator — Medical University of Lodz
Locations (1):
- Oddział Kliniczny Gastroenterologii Ogólnej i Onkologicznej USK nr 1 im. N. Barlickiego w Łodzi, Lodz, Poland

IPD SHARING:
Plan to Share IPD: No